CLINICAL TRIAL: NCT06510660
Title: Adebrelimab with or Without Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Prospective, Phase 2 Trial
Brief Title: Adebrelimab ±Induction Chemotherapy Followed by Concurrent Chemoradiotherapy for Unresectable Locally Advanced ESCC
Acronym: RICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yong Yang, principal investigator, Fujian Medical University Union Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RICE
Record Dates: First submitted 2024-04-01; First posted 2024-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma; Immunotherapy; Biomarkers
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adebrelimab+Sequential Concurrent Chemoradiotherapy (Experimental): Participants with CPS score ≥10 were enrolled.
  Induction therapy: adebrelimab 1200mg iv d1 q3w x 2 cycles for 6 weeks.
  Concurrent chemoradiotherapy: carboplatin AUC=2 / cisplatin 25mg/m2 d1 qw + paclitaxel 50mg/m2 / nab-paclitaxel 60mg/m2 d1 qw for a total of 5 weeks; radiotherapy:50Gy/25f, completed in 5 weeks.
  Interventions: Drug: adebrelimab
- Adebrelimab+Chemotherapy+Sequential Concurrent Chemoradiotherapy (Experimental): Participants with CPS score <10 were enrolled.
  Induction therapy: adebrelimab 1200mg iv d1 q3w + carboplatin AUC=6 / cisplatin 75mg/m2 d1 q3w + paclitaxel 175mg/m2 / nab-paclitaxel 260mg/m2 d1 q3w × 2 cycles for 6 weeks.
  Concurrent chemoradiotherapy: carboplatin AUC=2 / cisplatin 25mg/m2 d1 qw + paclitaxel 50mg/m2 / nab-paclitaxel 60mg/m2 d1 qw for a total of 5 weeks; radiotherapy:50Gy/25f, completed in 5 weeks.
  Interventions: Drug: adebrelimab

INTERVENTIONS:
Drug: adebrelimab — The study was divided into two cohorts based on CPS score, with those with CPS scores ≥10 receiving induction therapy with adebrelimab alone and those with CPS scores <10 receiving induction therapy with adebrelimab in combination with chemotherapy. At the end of the induction period, concurrent radiotherapy treatment was administered

SUMMARY:
To evaluate the efficacy and safety of adebrelimab with or without induction chemotherapy followed by concurrent chemoradiotherapy for unresectable locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This is a prospective, two-cohort, multicenter clinical study. Subjects received different treatments based on their CPS scores. During induction therapy, subjects in cohort 1 (CPS score ≥10) received adebrelimab, while cohort 2 (CPS score < 10) were administered adebrelizumab + carboplatin/cisplatin + paclitaxel/nab-paclitaxel. Both groups received carboplatin/cisplatin + paclitaxel/nab-paclitaxel combined radiotherapy during concurrent chemoradiotherapy. The primary endpoint was cCR rate.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, male or female;
2. Have not received systemic or localized treatment in the past;
3. Histologically or cytologically confirmed esophageal squamous cell carcinoma (AJCC 8th edition clinical stage II-IVA). IVB stage thoracic esophageal cancer with supraclavicular lymph node metastasis only. No surgical resection or refusal of surgical resection;
4. ECOG score of 0-1;
5. Life expectancy ≥ 3 months;
6. Adequate organ function;
7. Fertile men and women must agree to use contraception during the study period and for six months after the last drug used in the study；
8. Subjects will voluntarily enroll in the study, sign an informed consent form, be compliant, and cooperate with follow-up visits.

Exclusion Criteria:

1. Subjects with low body weight (BMI <18.5kg/m2) or ≥10% weight loss in the 2 months prior to screening;
2. Esophageal lesions with significant invasion of neighboring organs (e.g., aorta, trachea), or deep and large ulcers with a high risk of bleeding or fistula formation, or previous esophageal perforation or fistula within 6 months prior to screening;
3. Prior treatment with immunotherapy;
4. Treatment with any other clinical investigational drug or participation in another interventional clinical study within 4 weeks prior to first use of study drug;
5. Planning to receive or have received a prophylactic or live attenuated vaccine within 4 weeks prior to the first dose of study drug;
6. Receiving corticosteroid hormone therapy within 2 weeks prior to first use of study drug;
7. Subjects who have received a previous tissue/organ transplant or allogeneic hematopoietic stem cell transplant;
8. Active, known or suspected autoimmune disease;
9. Uncontrolled cardiac clinical symptoms or disease;
10. Active or uncontrolled serious infection (≥ CTCAE grade 2 infection);
11. Subjects with active tuberculosis or a history of active tuberculosis infection within 12 months prior to screening, with or without treatment;
12. History of interstitial lung disease (except radiation pneumonitis not treated with hormonal therapy), or history of non-infectious pneumonia;
13. Active hepatitis B virus or hepatitis C virus infection. Positive HIV test or known acquired immunodeficiency syndrome (AIDS);
14. Prior history of other malignancies within 5 years (except non-melanoma skin cancer, limited prostate cancer, or any early stage tumor treated by radical resection);
15. Known hypersensitivity to any of the investigational drugs or excipients;
16. The presence of other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the results of the study, and subjects who, in the opinion of the investigator, are unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
cCR | Up to 6 months.
  Clinical complete response rates.

SECONDARY OUTCOMES:
OS | From date of enrollment until the date of death from any cause, assessed up to 5 years.
  Overall survival.
PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  Progression free survival.
ORR | Up to 6 months.
  Objective response rate.
DoR | Up to 3 years.
  During of response.
DCR | Up to 6 months.
  Disease control rate.
Completion rate of concurrent radiotherapy | Up to 6 months.
  Calculate the percentage of patients who have completed concurrent radiochemotherapy.
AE | Up to 6 months.
  Adverse event,

OTHER OUTCOMES:
Biomarker analysis | Up to 6 months.
  Single-cell sequencing, whole-exome sequencing to screen effective biomarkers and explore their correlation with prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yang, Doctor, Principal Investigator — Fujian Medical University Union Hospital; Lei Zhao, Principal Investigator — Sun Yat-sen University
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No